CLINICAL TRIAL: NCT04334733
Title: The Impact of Preprocedural Informative Animation Display About Echocardiography and Intraprocedural Kaleidoscope Display on Anxiety in Children
Brief Title: The Impact of Preprocedural Animation About Echocardiography Display and Kaleidoscope Display on Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Collaborators: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Birsel Molu, PhD, Research assistant, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018/13 Osmangazi University
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Anxiety; Child, Only; Echocardiography
Keywords: Child; Anxiety; Echocardiography; Cartoon; Kaleidoscope
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This randomized controlled experimental study was carried out with 164 children in the 5-12 age group in the pediatric echocardiography unit of a Training and Research Hospital between February 2019 and November 2018. In the study, nonpharmacological methods were applied to the children in the experimental groups (Cartoon Group (n=41), Kaleidoscope Group (n=41), Cartoon+Kaleidoscope Group (n=41), Control group (Routine echocardiography) (41) . The data were collected using the "Introductory Information Form", "Children's Fear and Anxiety Scale (CFAS)".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cartoon group (Experimental): The children in the groups were distracted by watching cartoon 5 minutes before echocardiography.
  Interventions: Other: Cartoon group
- Kaleidoscope group (Experimental): The children in the groups were distracted by kaleidoscope during the echocardiography process, until the process was over.
  Interventions: Other: Kaleidoscope group
- Cartoon+Kaleidoscope group (Experimental): The children in the groups were distracted by watching cartoon 5 minutes before echocardiography and the children in the groups were distracted by kaleidoscope during the echocardiography process, until the process was over.
  Interventions: Other: Cartoon+Kaleidoscope group
- Control group (Experimental): No intervention was made to children in the control group
  Interventions: Other: Cartoon group; Other: Kaleidoscope group; Other: Cartoon+Kaleidoscope group

INTERVENTIONS:
Other: Cartoon group — The children in the groups were distracted by watching cartoon 5 minutes before echocardiography process.
  Arms: Cartoon group; Control group
Other: Kaleidoscope group — The children in the groups were distracted by kaleidoscope during echocardiography, until the process was over.
  Arms: Control group; Kaleidoscope group
Other: Cartoon+Kaleidoscope group — The children in the groups were distracted by watching cartoon 5 minutes before echocardiography process and then the children in the groups were distracted by kaleidoscope during echocardiography, until the process was over.
  Arms: Cartoon+Kaleidoscope group; Control group

SUMMARY:
Objective: The study was conducted for the purpose of determining the effect of making children aged 5 to 12 years watch a cartoon about echocardiography (ECO) procedure before the procedure and kaleidoscope during the procedure on their anxiety.

Material and Method: It is a randomized controlled study. The study was completed with a total of 164 children who came to have an ECO and met the sample selection criteria. There were four groups in the study which were as follows; the group that was made watch a cartoon about the procedure before the procedure, the group that was made watch a kaleidoscope during the procedure, the group that was made watch a cartoon about the procedure before the procedure and a kaleidoscope during the procedure and the control group in which routine applications of clinic were carried out.

Results: At the end of the study, it was determined that anxiety scores of the cartoon group, cartoon+kaleidoscope group and the kaleidoscope group were lower during the procedure than before the procedure (p<0,001). In the control group, it was determined that there was no significant difference between the anxiety scores before and during the procedure (p>0,05).

DETAILED DESCRIPTION:
The study was conducted for the purpose of determining the effect of making children aged 5 to 12 years watch a cartoon about echocardiography (ECO) procedure before the procedure and kaleidoscope during the procedure on their anxiety. It is a randomized controlled study. The study was conducted in the Pediatric Cardiology Polyclinic of Afyon Kocatepe University Ahmet Necdet Sezer Research and Application Hospital in the Province of Afyonkarahisar between 6 November 2018-1 February 2019. The study was completed with a total of 164 children who came to have an ECO and met the sample selection criteria. There were four groups in the study which were as follows; the group that was made watch a cartoon about the procedure before the procedure, the group that was made watch a kaleidoscope during the procedure, the group that was made watch a cartoon about the procedure before the procedure and a kaleidoscope during the procedure and the control group in which routine applications of clinic were carried out. Samples were assigned to the groups using permutation block randomization method. In order to collect data, an Introductory Information Form and the Child Fear Scale were used. The data acquired from the study were evaluated using the IBM SPSS Statistics 24 (Statistical Package for Social Sciences) package software. In our study, the experimental and control group children were found to be similar in terms of introductory characteristics (age, gender, educational level, family structure, number of children in family, illness and hospital experiences, information about ECO). At the end of the study, it was determined that anxiety scores of the cartoon group, cartoon+kaleidoscope group and the kaleidoscope group were lower during the procedure than before the procedure (p<0,001). In the control group, it was determined that there was no significant difference between the anxiety scores before and during the procedure (p>0,05).

ELIGIBILITY:
Inclusion Criteria:

* being healthy
* ability to express himself/herself verbally
* no sedation taken in the last eight hours
* having no visual or auditory problems
* Ecocardiography process is to be held for the first time

Exclusion Criteria:

* chronic disease
* mental disease
* neurological disease

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Female,Male
Enrollment: 164 (Actual)
Dates: Start 2018-10-06 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-12-25 (Actual)

PRIMARY OUTCOMES:
Children Fear Scale | 1 minute
  The Children Fear Scale was used to evaluate the children's fear and anxiety. Children Fear Scale is a 0-4 scale, showing five faces that range from a neutral expression (0 = no anxiety) to a frightened face (4 = severe anxiety). Preprocedural and procedural anxiety were evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Selçuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No